CLINICAL TRIAL: NCT05681871
Title: A South African Multi-centre Pilot Trial to Assess the Feasibility and Clinical Efficacy of Preoperative Oral Iron to Treat Preoperative Iron-deficiency Anaemia in Children Undergoing Elective Noncardiac Surgery
Brief Title: South African Paediatric Surgical Outcomes Study 2
Acronym: SAPSOS2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of Stellenbosch (Other); University of KwaZulu (Other)
Responsible Party: Principal Investigator, Heidi Meyer, Principal Investigator, Specialist Anaesthetist, Division of Paediatric Anaesthesia, Department of Anaesthesia & Perioperative Medicine, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N20221001
Record Dates: First submitted 2023-01-03; First posted 2023-01-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Paediatric Surgery; Anaemia; Iron Deficiency Anemia; Iron; Prospective Studies; Interventional Studies
Keywords: SAPSOS2
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — ferrous fumarate; Folic Acid

STUDY DESIGN:
Intervention Model Description: Prospective interventional quasi-experimental pre-post study South African multi-centre
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iron-deficiency anaemia (Experimental): Participants will receive oral iron supplementation for a minimum of 4 weeks prior to surgery
  Interventions: Dietary Supplement: Ferrous gluconate syrup or ferrous fumarate/folic acid tablets

INTERVENTIONS:
Dietary Supplement: Ferrous gluconate syrup or ferrous fumarate/folic acid tablets — Oral iron supplementation dosed based on body weight

SUMMARY:
Preoperative anaemia has been shown to be associated with worse outcomes after surgery in both adults and children. Limited research has been done on how common preoperative iron-deficiency anaemia (IDA) is in children and how best to treat it. Oral iron is a relatively cost-effective treatment for IDA. This study aims to show whether giving children with IDA oral iron for 6-12 weeks before their surgery significantly improves their haemoglobin.

DETAILED DESCRIPTION:
Studies in both paediatric and adult patients have shown an association between preoperative anaemia and increased postoperative morbidity and mortality, and transfusion rates. The incidence of preoperative anaemia in the secondary analysis of the SAPSOS cohort of children who underwent noncardiac surgery was 46.2%. IDA has been shown to represent up to 30% of preoperative anaemia in adults. Iron deficiency and IDA are of even greater concern in children, because of the negative impact it may have on cognitive performance.

A recent Cochrane review on the role of preoperative iron in reducing perioperative blood transfusion in adult patients found no significant reduction in the administration of allogeneic blood transfusion in patients who had received preoperative iron compared with those who did not. These findings were supported by the Preoperative intravenous iron to treat anaemia before major abdominal surgery (PREVENTT) trial which found no difference in blood transfusion or death between the patients who did and did not receive intravenous iron. However, these findings have generated much discussion in the literature and concerns have been raised about the clinical application of this study. The mean haemoglobin (Hb) difference between the two groups post intervention (0.47g.dl-1) highlights the need for greater understanding of the impact of an intervention on the absolute or relative increase in Hb when designing trials looking at the impact of iron treatment on perioperative outcomes. Dosing regimens of preoperative oral iron varies widely between studies further complicating the ability to draw conclusions of the role of oral iron in the treatment of preoperative anaemia.

In contrast with the findings of the Cochrane review and the PREVENTT trial, a meta-analysis of patient blood management programme (PBM) studies, many of which include preoperative iron treatment as a component, found that there was a reduction in exposure to red cell transfusions. Although, the meta-analysis also found the implementation of PBM was not associated with a reduction on in-hospital mortality or 30-day mortality, there was no additive benefit from multiple interventions and no trial showed that PBM were cost-effective. Not included in this meta-analysis were recently published studies on the implementation of preoperative anaemia screening clinics in adults in elective colorectal surgery and major surgery which demonstrated reductions in red cell transfusions, length of stay, and net costs in patients with IDA who were treated with preoperative intravenous iron. Similarly, a large study from Western Australia reported significant reductions in cost associated with the use of blood products, and improved patient outcomes, after implementation of a PBM.

Studies investigating the impact of increasing preoperative Hb on perioperative outcomes in children are primarily focused on blood loss and blood transfusion rates in surgery in which significant bleeding and frequent blood transfusion are anticipated and most of the children in these studies received preoperative erythopoeitin. The impact of preoperative oral iron as a stand-alone intervention to increases preoperative Hb are limited to 2 studies. A single retrospective study has reported on the impact of the introduction of preoperative oral iron without erythropoeitin (EPO) in children undergoing spinal surgery. They found a significant difference in intraoperative transfusion rates in patients who received a longer duration of preoperative oral iron therapy. The major limitation of the study was a lack of preintervention Hb, precluding the ability to assess the effect of iron supplementation on delta Hb. A subsequent study reviewing the impact of preoperative oral iron in paediatric cardiac patients found that iron supplementation resulted in an increase in preoperative Hb levels which was associated with reduced red blood cell transfusion volumes.

Given the high incidence of preoperative anaemia in children having surgery in South Africa in the public sector and its association with poorer postoperative outcomes, it is important to assess the feasibility of a pragmatic intervention to treat preoperative anaemia in the context of a resource-constrained setting. Although intravenous iron in combination with EPO may be more effective and have fewer side effects, oral iron is relatively inexpensive and widely available in South Africa. Regular deworming may also play an important role in the treatment of preoperative anaemia and has been shown to be an effective intervention to increase baseline Hb in school age children from low- and middle- income countries. We hypothesise that the implementation of preoperative anaemia screening and treatment of anaemic patients with a minimum of 6 weeks supplementation with oral iron will have a clinically significant effect on increasing the Hb in patients with preoperative IDA.

STUDY OBJECTIVE To evaluate the efficacy of oral iron supplementation in children diagnosed with preoperative IDA undergoing noncardiac surgery.

STUDY DESIGN Pre and post- South African multi-centre interventional study of oral iron supplementation to treat IDA in paediatric patients (age >6 months and <16 years) admitted to participating hospitals undergoing elective non-cardiac surgery. The intention is to present a representative sample of paediatric surgical patients with preoperative anaemia. This study will run from January 2023 until July 2023.

ETHICS APPROVAL Ethics approval will be in place at each hospital site prior to recruitment of patients. Informed consent, and assent where appropriate, must be obtained for each participant enrolled in the study.

IMPORTANCE OF STUDY Preoperative anaemia is associated with significant morbidity and mortality. The information gained from this study will contribute to a greater understanding of the incidence of preoperative IDA in children in South Africa and give insight into the feasibility and efficacy of oral iron supplementation to treat preoperative IDA.

ELIGIBILITY:
Inclusion Criteria:

* Age > 6 months to <16 years
* Noncardiac surgery
* Elective surgery
* Anaemic as per World Health Organisation criteria

Exclusion Criteria:

* Patient or parent refusal
* Unable to obtain written consent at the surgical outpatient clinic
* Surgery planned within 4 weeks from surgical outpatient visit
* Known history of acquired iron overload, family history of haemochromatosis or thalassemia
* Known reason for anaemia (e.g., untreated vitamin B12 or folate deficiency or haemoglobinopathy)
* Treatment with oral iron, erythropoietin, IV iron therapy or blood transfusion in the previous 12 weeks
* Known hypersensitivity to oral iron or other contraindication to oral iron
* Temperature > 38.0 °C or receiving non-prophylactic antibiotics
* Acute liver failure

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 755 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Delta Haemoglobin = Change in haemoglobin pre- and post- oral iron supplementation | 4-12 weeks
  g/dL

SECONDARY OUTCOMES:
Incidence of iron-deficiency anaemia | 24 months
  Incidence of iron-deficiency anaemia

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M Meyer, MBChB, Principal Investigator — University of CapeTown
Locations (2):
- South Africa (2):
  - Tygerberg Hospital, Cape Town, Western Cape
  - Red Cross War Memorial Children's Hospital, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Data sharing agreement has been finalised between the University of Cape Town and Professor Susan Goobie and Dr. Steven Staffa at Boston Children's Hospital. Purpose of this agreement is for statistical analysis and manuscript development. All shared data will undergo de-identification. Shared data includes eligibility, consent, reasons for exclusion, and de-identified record IDs, patient demographics, comorbidities, deworming status, planned date of surgery, hemocue results, pre-intervention formal Hb, MCV, reticulocyte count, CRP, ferritin levels, TSAT, information regarding medication compliance and any experienced side-effects, date of repeat Hb and post-intervention formal Hb, and serious adverse events.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact researchcontracts@uct.ac.za

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT05681871/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT05681871/ICF_001.pdf